CLINICAL TRIAL: NCT01089764
Title: A Randomized Controlled Trials of Couplelinks.ca: The First Online Couples Intervention for Young Women Dealing With Breast Cancer and Their Male Partners
Brief Title: Couplelinks.ca - An Online Intervention for Couples Affected by Breast Cancer
Acronym: couplelinks
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Canadian Breast Cancer Research Alliance (Other)
Collaborators: York University (Other); Sunnybrook Health Sciences Centre (Other); British Columbia Cancer Agency (Other); CancerCare Manitoba (Other); Queen Elizabeth II Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Karen Fergus, PhD, Canadian Breast Cancer Research Alliance
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H10-00300
Record Dates: First submitted 2010-03-17; First posted 2010-03-19 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-08

CONDITIONS: Distress; Breast Cancer; Depression; Anxiety
Keywords: breast neoplasm; breast cancer; behavioral intervention; online support; relationship distress; dyadic coping
MeSH Terms: conditions — Breast Neoplasms; Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Couplelinks.ca Intervention (Experimental): Intervention arm - Couple participates in the Couplelinks.ca program.
  Interventions: Behavioral: Couplelinks.ca website
- No Intervention (No Intervention): Couple is waitlisted for participation in the Couplelinks.ca program.

INTERVENTIONS:
Behavioral: Couplelinks.ca website — Participation in the Couplelinks.ca program, an online intervention.
  Other Names: Couplelinks.ca program
  Arms: Couplelinks.ca Intervention

SUMMARY:
Women diagnosed with breast cancer (BC) at or before the age of 50 experience more distress and poorer quality of life than women diagnosed later in life. Although adequate spousal support is a protective factor for women with BC, spouses are often unprepared to handle the myriad practical and emotional demands posed by the illness. Furthermore, despite the growing number of recommendations for couple interventions in relation to BC, traditional counselling approaches may fail to meet the needs of young couples who have unique concerns and tight constraints on their time. The proposed project addresses the void in the psycho-social support available to young couples via an innovative, online psychoeducational intervention tailored specifically to their needs.

DETAILED DESCRIPTION:
Couplelinks.ca is a custom-designed website offering a professionally facilitated, couple-centred intervention that entails informational, experiential, and interactive components. Six Dyadic Learning Modules (DLM) form the core of the program and are undertaken on a weekly basis.

A funded pilot study examining the feasibility and benefit of Couplelinks.ca utilized a non-randomized, pre-post test design to assess the process and outcomes of the intervention. Qualitative feedback also informed the evaluation. Preliminary findings were promising and provided justification for further evaluation of the program's effectiveness.

The current study is the next logical step: a larger-scale Phase III study to determine whether this BC-specific, relationship-enhancement program leads to improved relationship and psychological outcomes for young couples affected by BC. It is a randomized controlled trial (RCT) comparing level of distress and dyadic adjustment in couples who have participated in the Couplelinks.ca educational program to those who have not participated and were instead put on a wait-list for participation.

ELIGIBILITY:
Inclusion Criteria:

* couples where woman has received a diagnosis of nonmetastatic breast carcinoma;
* diagnosis was within the last 36 months;
* woman is age less than or equal to 50 at age of diagnosis;
* completed or are nearing the end of active treatment;
* couples must be in a committed, heterosexual relationship;
* fluent in English with the ability to read and write in English.

Exclusion Criteria:

* non-heterosexual couples;
* women older than 50;
* previous diagnosis of moderate to severe psychological problems that may interfere with capacity to benefit from the intervention;
* couples who plan to participate in couple counselling during the 5-month study duration.

Ages: 18 Years to 53 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 260 (Estimated)
Dates: Start 2010-11; Primary Completion 2015-05 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Revised Dyadic Adjustment Survey RDAS | T0= 0 weeks, T1= 8 weeks, T3= 3 months
  The Revised Dyadic Adjustment Survey (RDAS) is a brief version of the 33 question Dyadic Adjustment Survey that assesses relationship adjustment.
Dyadic Coping | T0= 0 weeks, T1= 8 weeks, T3= 3 months
  Dyadic Coping assesses the degree to which partners feel that their coping efforts are reciprocal

CONTACTS AND LOCATIONS:
Overall Officials: Karen Fergus, PhD, Principal Investigator — York University/Sunnybrook Health Sciences Centre (Odette Cancer Centre)
Locations (5):
- Canada (5):
  - British Columbia Cancer Agency Research Centre, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - York University, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

REFERENCES:
- [Derived] Fergus K, Ahmad S, McLeod DL, Stephen J, Gardner S, Pereira A, Warner E, Carter W. Couplelinks - an online intervention for young women with breast cancer and their male partners: study protocol for a randomized controlled trial. Trials. 2015 Jan 29;16:33. doi: 10.1186/s13063-014-0534-8. PMID 25630357